CLINICAL TRIAL: NCT01495351
Title: Phase I Study of ABT-888 in Combination With Bortezomib and Dexamethasone in Patients With Relapsed Refractory Myeloma
Brief Title: Study of ABT-888 in Combination With Bortezomib and Dexamethasone in Patients With Relapsed Refractory Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Tom Baker Cancer Centre (Other); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM11-01; E24055 (Other: CHREB- University of Calgary)
Record Dates: First submitted 2011-11-16; First posted 2011-12-20 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ABT-888/Bortezomib (Experimental): Patients will be on a treatment schedule including twice daily oral dosing for 14 days followed by 1 week rest in combination with standard dosing of Bortezomib and Dexamethasone in a 21 days cycle for a total of 14 cycles.
  Interventions: Drug: ABT-888/Bortezomib

INTERVENTIONS:
Drug: ABT-888/Bortezomib — ABT-888 is given orally (PO) twice daily (every 12 hours) for 14 days in a 21 days cycle. First dose to be given within 1 hour of Bortezomib on day 1. Planned starting dose is 20 mg PO every 12 hours. Starting dose escalation is planned until an MTD is reached.

SUMMARY:
The combination of PARP inhibitor (ABT-888) with a proteasome inhibitors (bortezomib) have demonstrated significant anti-myeloma effects in preclinical lab and animal studies. The goal of this phase I trial is to evaluate in patients with relapsed or refractory multiple myeloma the safety, toxicity profile and tolerability of ABT-888 (Veliparib) administered on a schedule including twice daily oral dosing for 14 days followed by 1 week rest in combination with standard dosing of Bortezomib.

DETAILED DESCRIPTION:
This is a dose-finding / dose escalation phase I trial of ABT-888 (Veliparib) in combination with Bortezomib and Dexamethasone in patients with relapsed or refractory multiple myeloma. ABT-888 is given orally (PO) twice daily (every 12 hours) for 14 days in a 21 days cycle.

First dose to be given within 1 hour of Bortezomib on day 1. Planned starting dose is 20 mg PO every 12 hours. Starting dose escalation is planned until an MTD is reached.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple myeloma.
* Measurable disease, according to the International Myeloma Working Group criteria.
* ECOG performance status 0, 1 or 2.
* Patients must have received prior treatment for MM and have relapsed or progressed on prior therapy; no limit on number of prior treatment regimens, but prior treatment must be completed 2 weeks prior to registration. Prior exposure to Bortezomib is not an exclusion criteria as long as patients did not progress or relapse while receiving or within 3 months of completing trt with bortezomib
* Prior radiation, completed at least 4 weeks prior to registration, is permitted.
* Adequate marrow reserve, liver and renal function

Exclusion Criteria:

* patients with a history of other malignancies, except: adequately treated nonmelanoma skin cancer, curatively treated in-situ cancer of the cervix, prostate cancer with stable PSA for > 3 years, or other solid tumours curatively treated with no evidence of disease for > 5 years.
* Patients with preexisting grade 2 (or higher) sensory neuropathy or grade 1 sensory neuropathy with neuropathic pain.
* Pregnant or lactating women
* Patients receiving concurrent treatment with other anti-cancer therapy any other investigational agents.
* Active or uncontrolled infections
* Patient with known documented congenital or acquired risk factor for thromboembolic event
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02-10 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) of ABT-888. | 21 Day Cycle
  Study follows a modified dose escalation scheme with a 3+3 design (3 to 6 patients per dose level or cohort). Only the ABT-888 dose will be escalated with a maximum dose of ABT-888 of 100 mg PO BID. If >1 out 6 patients at any dose level suffer dose limiting toxicity, then dose escalation is stopped, and this dose is declared as MTD. 3 additional patients will be entered at the next lowest dose level. The recommended phase 2 dose is defined as the dose level with ≤ 1 out of 6 patients experiencing DLTs at the highest dose level below the MTD.
Identify the Dose Limiting Toxicities (DLT) of ABT-888 | 21 Day Cycle
  All adverse events, including DLTs, are graded according to the NCI CTCAE, v4.0. A DLT is defined as any grade 3 or higher non-hematologic toxicity, or any grade 4 hematologic toxicity, considered by the investigator to be related to the study drugs and occurring during Days 1-22 of Cycle 1.

SECONDARY OUTCOMES:
Activity Objective - Preliminary assessment of the anti-tumor activity of ABT-888 | 21 day cycle
  Response to study drugs is assessed at the end of each cycle according to the International Myeloma Working Group (IMWG) response criteria.
Exploratory Objective - Preliminary assessment of potential biomarkers | 24 months
  Gene expression profiling is performed at baseline and compared between responders versus non-responders in order to identify a "treatment response signature". 2.5 mg of RNA will be extracted from plasma cells sorted from pre-treatment (D1, cycle 1) (n=20) and post-treatment (D11, cycle 1) (n=20) bone marrow aspirates collected from patients treated in the extension cohort. cRNAs will be hybridized onto the U133 Plus 2.0 gene chips and raw data files acquired using Affymetrix Microarray Suite version 5.1 software and analyzed with the Partek Genomics Suite v6.4.
Exploratory Objective - Determine in vivo the effect of ABT-888 on PARP inhibitors. | 24 Months
  Poly-ADP-ribose (PAR) levels are measured in sorted CD138+ plasma cells from pre-ABT-888 treatment on day 1 cycle1, as well as post ABT-888 treatment (within 4-6 hours) on days 4 and 11. PAR levels will be measured by standardized ELISA assays (HT PARP in vivo Pharmacodynamic Assay II™, Trevigen).
Determine invivo the effects of Bortezomib on the plasma cells DNA genes expression and function | 24 Months
  Gene expression profiling is performed at baseline prior to treatment with bortezomib and on days 4 and 11 post bortezomib treatment. 2.5 mg of RNA will be extracted from plasma cells sorted from bone marrow aspirates collected from patients treated on trial. cRNAs will be hybridized onto the U133 Plus 2.0 gene chips and raw data files acquired using Affymetrix Microarray Suite version 5.1 software and analyzed with the Partek Genomics Suite v6.4.

CONTACTS AND LOCATIONS:
Overall Officials: Nizar J Bahlis, M.D., Study Chair — Tom Baker Cancer Centre, University of Calgary
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada